CLINICAL TRIAL: NCT07027462
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Clinical Trial Of A Mushroom Blend To Evaluate Its Impacts On Gastrointestinal and Overall Quality Of Life and Microbiome Makeup In Healthy Adults
Brief Title: Effects of a Mushroom Blend on Gastrointestinal Symptoms and the Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: M2 Ingredients (Industry); Substantiation Sciences, LLC (Unknown)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00144162
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Gastrointestinal Discomfort; Mood; Mushroom

STUDY DESIGN:
Intervention Model Description: Between-subjects, placebo-controlled study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, the research team interacting with the participants, and the primary data analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will be consuming a blend of cordyceps, reishi, and lion's mane mushrooms .
  Interventions: Dietary Supplement: Mushroom blend
- Control (Placebo Comparator): Organic Acacia Gum will be the placebo product for this study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Mushroom blend — A mushroom blend that is targeted to improve gastrointestinal symptoms.
  Arms: Experimental
Other: Placebo — Placebo product.
  Arms: Control

SUMMARY:
This study will investigate the efficacy of a mushroom blend to improve gastrointestinal symptoms and mood. It will also be determining if the mushroom blend has an effect on the gut microbiome and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 30 to 60 years of age (inclusive).
* Subject has provided written and dated informed consent.
* Individual indicates they experience occasional GI discomfort, and have never been diagnosed with any gastrointestinal disorder, yet have occasional complaints of bowel irregularity, bloating or discomfort (after meals or beverages).
* Subject may express that they experience occasional after-snack or a meal, intestinal gas-related symptoms including abdominal discomfort, cramps, distended feeling/bloating, and or flatulence as part of the study entry criteria.
* Occasional GI distress will be defined as < 3 times per week over the prior 6 weeks, with each episode resolving within 24 hours and not requiring medical intervention.
* Body Mass Index (BMI) 19 to 34.9 kg/m2 (normal weight to class I obesity)
* Subject is a non-smoker.
* Subject agrees to not use any new vitamin, mineral, or other dietary supplement product until after study completion.
* Subject agrees to provide a stool sample for microbiota analysis per the study protocol.
* Subject is willing and able to comply with the protocol and the scheduled study visits.
* Subject will be asked about dietary supplementation use within the past 6 months.

  * If subject began taking a supplement within the past month, participant will be asked to discontinue supplement use followed by a 2-week washout prior to participation.
  * In all other cases, supplement use will be asked to be maintained throughout the study.

Exclusion Criteria:

* Subject has any of the following medical conditions:

  * Gastrointestinal disease or any GI diagnosed disorder (i.e., dyspepsia, functional dyspepsia, gastrointestinal reflux, etc.)
  * active heart disease
  * uncontrolled high blood pressure (≥ 140/90 mmHg)
  * renal or hepatic impairment/disease
  * Type I or II diabetes
  * bipolar disorder
  * Parkinson's disease
  * unstable thyroid disease
  * immune disorder (such as HIV/AIDS)
  * Any medical condition deemed exclusionary by the Principal Investigator (PI)
* Subject has a history of cancer (except localized skin cancer without metastases) within 5 years prior to screening.
* Subject is currently taking any blood thinners.
* Subject has a medical condition that is known to impact the gastrointestinal system and functions.
* Subject is currently taking or has within the prior 120 days any prescription antibiotics, or supplemental probiotic or prebiotics (30-day washout is acceptable).
* Subject is currently taking supplemental (OTC medicine or dietary supplements) of any laxative or bowel function stimulant [i.e., Ri-Mucil, Metamucil (psyllium), Colace, Milk of Magnesia, MiraLAX, FiberCon (polycarophil), DulcoLax, etc.]
* Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).
* Subject is taking a prescription medication deemed exclusionary by the Principal Investigator (PI).
* Subject has an allergy to any ingredients in the Study Product.
* Subject has a history of drug or alcohol abuse in the past 12 months.
* Subject has a history of a psychiatric illness or mental health disorder (including for drug or alcohol treatment) that required hospitalization in the prior 12 months.
* Subject has any condition or health history abnormality that in the expert opinion of the PI, participation in the study would compromise the safety of the subject or the quality of the study data.
* The subject is participating in or has participated in another clinical research study within 30 days prior to the Screening visit.
* Subject is consuming any of the study products already.
* Subject is diagnosed with a stress-disorder.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the gastrointestinal symptoms rating scale. | Visit 2 (Day 0), Visit 3 (Day 19-21), Visit 4 (Day 42)
  To determine if the study product has any effect on digestion. Scores range from 0 - 45, with higher scores indicating severe gastrointestinal issues.
Changes in Assessment of Constipation - Quality of Life | Visit 2 (Day 0), Visit 3 (Day 19-21), Visit 4 (Day 42)
  To determine if the study product has any effect on quality of life in individuals suffering from constipation. It is scored as means of each item, ranging from 0 - 4 with higher scores indicating worse quality of life.
Changes in total mood disturbances | Visit 2 (Day 0), Visit 3 (Day 19-21), Visit 4 (Day 42)
  To determine if the study product has any effect on mood states. The total mood is calculated by adding the negative subscales (tension, depression, fatigue, confusion, and anger) subtracting the positive subscales (vigor, esteem-related affect). Higher scores indicate worse moods.
Changes in the gastrointestinal microbiota alpha diversity | Visit 2 (Day 0) and Visit 4 (Day 42)
  To determine if the study product has any effect on the gut microbiota composition.
  6S rRNA gene (V4 amplicon) sequencing will be performed to profile the gut microbial community of frozen fecal samples collected from all humans to ascertain how the Mushroom Blend impacts gut microbial community structure of alpha diversity.
Changes in the gastrointestinal microbiota beta diversity | Visit 2 (Day 0) and Visit 4 (Day 42)
  To determine if the study product has any effect on the gut microbiota composition.
  6S rRNA gene (V4 amplicon) sequencing will be performed to profile the gut microbial community of frozen fecal samples collected from all humans to ascertain how the Mushroom Blend impacts gut microbial community structure of beta diversity.
Changes in the gastrointestinal microbiota relative abundance of specific gut bacteria based on amplicon sequence variants. | Visit 2 (Day 0) and Visit 4 (Day 42)
  To determine if the study product leads to an increase or decrease in the gastrointestinal microbiota relative abundance of specific gut bacteria. 6S rRNA gene (V4 amplicon) sequencing will be performed to profile the gut microbial community of frozen fecal samples collected from all humans to ascertain how the Mushroom Blend impacts gut microbial relative abundance of specific gut bacteria based on amplicon sequence variants.
Changes in water-soluble polar metabolites. | Visit 2 (Day 0) and Visit 4 (Day 42)
  To determine if the study product leads to an increase or decrease in water-soluble polar metabolites. positive and negative metabolites will be extracted from serum using a protocol optimized for water soluble polar metabolite analysis using Liquid Chromatography coupled with Mass Spectrometry (LC-MS).

SECONDARY OUTCOMES:
Frequency of gastrointestinal distress. | Baseline and Day 42.
  To determine if the study product reduces the frequency of reported gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No